CLINICAL TRIAL: NCT05427552
Title: Exploring the Cortical Hemodynamic Response of Excitatory Brain Stimulation: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HSEARS20200120005-01
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Theta-Burst stimulation (iTBS); Functional near-infrared spectroscopy (fNIRS); Concurrent TMS/fNIRS; Prefrontal hemodynamic response
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Healthy volunteers will receive iTBS three times with three different intensities separated by one week to investigate the prefrontal hemodynamic response to different stimulation intensities.
Who Masked: Participant
Masking Description: Participants will not be informed of the stimulation intensities.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Prefrontal hemodynamic response to 50% rMT iTBS (Experimental): Participants will receive 50% rMT iTBS over left DLPFC in this arm. The prefrontal hemodynamic response will be observed simultaneously before, during, and after iTBS using fNIRS.
  Interventions: Device: Intermittent theta-burst stimulation (iTBS)
- Prefrontal hemodynamic response to 70% rMT iTBS (Experimental): Participants will receive 70% rMT iTBS over left DLPFC in this arm. The prefrontal hemodynamic response will be observed simultaneously before, during, and after iTBS using fNIRS.
  Interventions: Device: Intermittent theta-burst stimulation (iTBS)
- Prefrontal hemodynamic response to 90% rMT iTBS (Experimental): Participants will receive 90% rMT iTBS over left DLPFC in this arm. The prefrontal hemodynamic response will be observed simultaneously before, during, and after iTBS using fNIRS.
  Interventions: Device: Intermittent theta-burst stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent theta-burst stimulation (iTBS) — The iTBS will be applied over lDLPFC with three different intensities. The investigators put the NIRS probe under the TMS coil to detect the hemodynamic signal simultaneously, and the applied rMT was adjusted based on Stokes et al., 2007. The equation is AdjMT% = MT + 2.8 * (Dsitex - Dm1), and the thickness of the probe is 6mm, therefore, 2.8*6=16.8(%) were added to the normal intensity.
  Other Names: Transcranial magnetic stimulation (TMS)

SUMMARY:
Intermittent theta-burst stimulation (iTBS) is a promising treatment for major depressive disorder. However, fewer than 50% of patients show sufficient response. Therefore, the optimal treatment protocol is worth investigating. Recent studies show that the relationship between stimulation intensity and prefrontal hemodynamic response is not linear but in an inverse U-shape by exploring the hemodynamic changes before and after iTBS. Concurrent transcranial magnetic stimulation (TMS)/functional near-infrared spectroscopy (fNIRS) setup allows the investigators to observe the prefrontal hemodynamic response during stimulation.

The aim of this study is to investigate the effects of different intensities on brain activity during and after the stimulation using fNIRS.

DETAILED DESCRIPTION:
Please refer to the full proposal

ELIGIBILITY:
Inclusion Criteria:

* Right-handed

Exclusion Criteria:

* history of epilepsy, seizures, or convulsions
* current or past diagnosis of neurological disorders, such as head injuries, strokes, encephalitis, epilepsy, Parkinson's, or Alzheimer's
* current or past diagnosis of psychiatric disorders, such as depression, anxiety, schizophrenia, or autism
* with metal implants, such as a cochlear implant, neurostimulator, or cardiac pacemaker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Oxygenated hemoglobin (HbO) change compared to baseline | During and post TBS-fNIRS measurement, up to 3 months
  iTBS-induced HbO change in the DLPFC before, during and after stimulation

SECONDARY OUTCOMES:
Deoxygenated hemoglobin (HbR) Change compared to baseline | During and post TBS-fNIRS measurement, up to 3 months
  iTBS-induced HbR change in the DLPFC before, during and after stimulation
Oxygen saturation change compared to baseline | During and post TBS-fNIRS measurement, up to 3 months
  iTBS-induced oxygen saturation change in the DLPFC before, during and after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Georg S Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No